CLINICAL TRIAL: NCT03223987
Title: Influence of a Food Supplement on the Gut Microbiome in Healthy Obese Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bio-Strath AG (Industry)
Collaborators: Zentrum für Adipositas- und Stoffwechselmedizin Winterthur GmbH (Industry)
Responsible Party: Principal Investigator, Peter Joller, PhD, Peter Joller, PhD Clinical Immunology FAMH, Bio-Strath AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BS2016.1
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Overweight
Keywords: 16S rRNA; Microbiome; Strath Herbal Yeast Preparation
MeSH Terms: conditions — Overweight | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Before-after intervention, open label study
Masking Description: First letter of prename, second and third letter of name.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): The study is one armed
  Interventions: Dietary Supplement: Strath® Kräuterhefe Original (liquid)

INTERVENTIONS:
Dietary Supplement: Strath® Kräuterhefe Original (liquid) — The food supplement is taken 3 x 1 coffee spoon à 5ml = 15ml per day for three weeks.
  Stool analysis at 2nd visit and last visit. Before-after study.

SUMMARY:
Before and after study in obese women 25-35 years old, BMI 30-35, taking Strath® Kräuterhefe Original (liquid), Herbal Yeast Food Supplement for three weeks. At the beginning and after three weeks of the study a stool sample is provided. These samples are analysed with 16S rRNA analysis down to species level.The results are interpreted with the PICRUSt classification and Alpha Diversity Analysis and compared to internationally accepted data bases.

DETAILED DESCRIPTION:
Intervention: Variation of the gut microbiome via intake of an herbal yeast preparation.

Participants: healthy obese women between 25 and 35 years. Intervention to be studied: Intake of Strath® Kräuterhefe Original (liquid), Herbal Yeast Food Supplement over 3 weeks, stool analysis.

Sequence and duration of all study periods: 7 weeks per proband.

Week -4 - -2: Pre-Phase Hand out study information First check of inclusion/exclusion criteria

Week -2: Initiation-Phase Signed "Informed Consent" Second check of inclusion/exclusion criteria Complete assessment Part I, II (see 8.2) Start assessment Part IV (see 8.2)

Week 0: Intervention-Phase Implementation of food supplement Complete assessment Part III (see 8.2) Third check of inclusion/exclusion criteria

Week 3: Evaluation-Phase Complete assessment Part II, III and IV Fourth check of inclusion/exclusion criteria Compliance control

5.2 Methods of minimising bias (ICH/E6 6.4.3; AGEK 4.3; SPIRIT #16, 17) ICH: A description of the measures taken to minimize/avoid bias, including: Randomization, Blinding.

Homogenous sample selection. 5.2.1 Randomisation Not applicable

5.2.2 Blinding procedures Not applicable

5.2.3 Other methods of minimising bias The investigators are going to do a semi-quantitative screening to determine a participant's nutritional habits.

Questions about their nutritional habits asked in the screening (via questionnaire);

1. Does the participant have a particular or alternative lifestyle (e.g. vegan, vegetarian, only eating raw fruits and vegetables, etc.)?

   - if yes → excluded
2. Does the participant control your nutrition in any form (food diary, app, counting calories, etc.)?

   - if yes → excluded
3. Does the participant consciously eat food to strengthen your immune system or do you take additional supplements to influence your intestinal bacteria (e.g. pro- and/or prebiotic food like Actimel, Activia, etc.)?

   - if daily or weekly → excluded
4. Does the participant exercise regularly? If yes, how often? - if 3h/week or more → excluded
5. On how many days per week does the participant eat meat or meat products?

   - if less then twice and more than five times peer week → excluded
6. On how many days per week does the participant eat fish?

   - if less or more than twice per week / 5 times per month → excluded
7. On how many days per week does the participant eat salad, vegetables or vegetable juice (not counting potatoes)?

   - if less than 5 days per week → excluded
8. On how many days per week does the participant eat fruits or drink fruit juices approximately?

   - if less than 5 days per week → excluded
9. On how many days per week does the participant drink or eat milk or milk products approximately? - if less than 4 days per week → excluded

ELIGIBILITY:
Inclusion Criteria:

* Women, 25 to 35 years, BMI 30-35
* German speaking
* Smartphone owner

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* any kind of nutritional intervention due to a disease in the past 6 months
* any mean of weight reduction in the past 6 months
* Severe health problems in the last 6 months
* Chronic digestive system problems
* Medication against constipation and diarrhea
* Mental problems
* Major surgery
* Allergies or Atopy
* Drug intolerance
* Antibiotics within 12 months before study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — xx genome
Enrollment: 26 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Quantitative difference in microbiome composition. | Six weeks.
  BoosterShot shotgun sequencing analysis down to the species level and compared with internationally accepted data banks. Comparison before-after.

SECONDARY OUTCOMES:
BMI | Three weeks
  Analysing the influence of the food additive on obesity parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Joller, PhD, Study Director — Dr.Joller BioMedical Consulting
Locations (1):
- Center for Obesity and Metabolism Adimed - Zentrum für Adipositas- und Stoffwechselmedizin Winterthur GmbH Lagerhausstrasse 9, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
After study termination we decide if for publication other researchers will be involved